CLINICAL TRIAL: NCT07103915
Title: Patient Satisfaction and the Effectiveness of Intranasal Lidocaine Spray Versus Nasogastric Tube Administration in the Emergency Room
Brief Title: Intranasal Lidocaine Spray Versus Nasogastric Tube Administration in the Emergency Room
Acronym: Lidocaine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Alp Şener, Associate professor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: No:E1-23-3927
Record Dates: First submitted 2025-07-25; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Nasogasrtic Tube Insertion
Keywords: intranasal lidocaine; numeric rating scale; Pain; Lidocaine spray; nasogastric tube
MeSH Terms: conditions — Pain | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: prospective, randomized, placebo-controlled, double-blind study, single centered
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- %10 lidocaine spray (Experimental): Drug: Lidocaine 10% Spray Two sprays in each nostril administered 1 minute prior to NGT insertion
  Interventions: Drug: Lidocaine 10% Spray
- Placebo (Placebo Comparator): Drug: Placebo Spray (Ethanol-matched solution without lidocaine)
  Two sprays in each nostril, same protocol
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lidocaine 10% Spray — This study evaluates whether intranasal 10% lidocaine spray reduces pain and improves first-pass success during nasogastric tube (NGT) insertion compared to placebo.
  Other Names: Xylocaine nasal spray
  Arms: %10 lidocaine spray
Other: Placebo — Drug: Placebo Spray (Ethanol-matched solution without lidocaine)
  Other Names: Placebo nasal spray
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate whether 10% intranasal lidocaine spray reduces pain and improves the success rate of nasogastric tube (NGT) insertion compared to placebo in adult emergency department patients.

The study's primary outcomes were:

Procedure success rate (first-pass success)

Pain during insertion, measured by the Numeric Rating Scale (NRS), where 0 = "no pain" and 10 = "worst possible pain".

The secondary outcomes included:

Duration of the procedure (in seconds)

Overall success rate (eventual successful insertion regardless of attempts)

Pain score at the 5th minute post-procedure (NRS)

Patient preference for the same method in future procedures (yes/no)

Procedure satisfaction, assessed using an NRS-based score from 0 ("not satisfied at all") to 10 ("completely satisfied").

Participants were randomized to receive either lidocaine or placebo spray intranasally before standard NGT insertion. Pain, success rate, and satisfaction were compared between groups.

DETAILED DESCRIPTION:
This randomized controlled trial aims to evaluate the effect of intranasal lidocaine 10% spray on patient comfort and pain during nasogastric tube (NGT) insertion in the emergency department. NGT placement is often associated with significant discomfort and anxiety, which can reduce procedural success and patient cooperation.

Eligible adult patients requiring nasogastric tube insertion in the emergency setting will be randomly assigned to receive either intranasal lidocaine spray or a placebo spray prior to the procedure. Both groups will undergo standard NGT placement performed by emergency physicians.

The primary outcome of the study is the level of pain experienced during the procedure, assessed using the Visual Analog Scale (VAS). Secondary outcomes include patient satisfaction, ease of tube placement from the clinician's perspective, vital signs during the procedure, and any adverse effects related to the spray or procedure.

The study seeks to determine whether intranasal lidocaine spray improves procedural comfort and increases overall satisfaction during a commonly performed yet unpleasant emergency intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Presentation to the emergency department during the study period and research assistant's working hours
* Clinical indication for nasogastric tube (NGT) insertion, including:
* Ileus
* Gastrointestinal bleeding monitoring
* Oral feeding difficulties due to neurological or similar disorders
* Intoxication
* Provided written informed consent
* Did not meet any of the exclusion criteria

Exclusion Criteria:

* Hemodynamic instability (hypotension, tachycardia, tachypnea, or hypoxia)
* Cognitive impairment or inability to cooperate
* Hearing or visual impairment
* Inability to sit upright
* History of epistaxis
* Use of anticoagulant medication
* Coagulopathy (elevated PT/aPTT or thrombocytopenia)
* Increased risk of aspiration
* Known lidocaine allergy
* History of arrhythmia, cardiac disease, or cardiac arrest
* Pregnancy
* Nasopharyngeal obstructive pathology
* Facial or nasal trauma preventing NGT insertion
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
First-Pass Success Rate | During initial NGT insertion attempt
  Rate of initial procedure success
Insertion pain score | During nasogastric tube insertion
  Numerical Rating Scale:Level of pain experienced during nasogastric tube insertion, as reported by the patient using the Numerical Rating Scale (NRS). The NRS is a validated 10-point scale ranging from 1 (no pain) to 10 (worst imaginable pain). Higher scores reflect more intense pain perception.

SECONDARY OUTCOMES:
Nasogastric tube insertion time | During procedure (in seconds)
  Evaluation of nasogastric tube insertion time with/without Lidocaine spray
Patient satisfaction | Immediately after procedure
  Patient preference for the subsequent attempts:Patient satisfaction will be evaluated immediately after the procedure by asking the participant which method they would prefer if a nasogastric tube were needed again. Preference will be recorded as an indicator of satisfaction. The unit of measure is "patient-reported preference (yes/no)." Higher willingness to repeat the same method is interpreted as higher satisfaction.
Pain Score at 5 Minutes | 5 minutes after completion of insertion
  Measured on the same Numeric Rating Scale(NRS):Pain intensity will be assessed using the Numeric Rating Scale (NRS), a validated tool ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst possible pain. The score will be recorded 5 minutes after the completion of the insertion procedure. Higher scores correspond to greater pain intensity.
Overall Procedure Success | Within 5 minutes of placement
  Successful NGT placement, regardless of number of attempts.

CONTACTS AND LOCATIONS:
Overall Officials: Kadir Yenal, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital Emergency Medicine Department, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared upon reasonable request by journal editors.
Supporting Information: Study Protocol, SAP
Time Frame: Individual participant data and supporting information will be available throughout the publication process, from August 15, 2024 to August 15, 2026.
Access Criteria: Access to individual participant data and supporting information will be granted to qualified researchers who submit a reasonable request, including a detailed research proposal. Approved researchers will be able to access anonymized datasets and relevant documentation via a secure data-sharing platform following approval by the study's data access committee.